CLINICAL TRIAL: NCT04748250
Title: Effect of Soy Phytoestrogens and Acupuncture on Bone Mineral Density in Female Athlete Triad at Adolescence Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hend Reda Sakr (Other)
Responsible Party: Sponsor-Investigator, Hend Reda Sakr, Principal investigator and Lecturer at Department of Physical Therapy for Woman's Health, Badr University
Organization: Badr University (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Hend1
Record Dates: First submitted 2021-02-04; First posted 2021-02-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Osteoporosis, Osteopenia
Keywords: female athlete triad
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Female Athlete Triad Syndrome | interventions — Soybean Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupuncture Group (Experimental): This group will receive acupuncture therapy for 30 minutes, three times per week for six months using the internationally recognized standard acupuncture needle which is 3 cm long with diameter o.3 mm, pushing it with twisting movement to the required depth until the De Qi sensation will be obtained.
  Interventions: Device: Acupuncture needles
- Soy Group (Experimental): This group will receive soy products for six months which including: Soy milk: 100 millilitre of soy milk every day, every bottle of original soy milk contains 300 millilitre or Soy beans: 100 gram of cooked soy beans per day.
  Interventions: Dietary Supplement: Soy phytoestrogens
- Acupuncture and Soy Group (Experimental): Every patient in this group will receive acupuncture therapy sessions in abdominal acu-points as in group (A) for 30 minutes, three times per week for six months in addition to administration of soy products in the form of soy milk or soy beans daily in breakfast for three months as in group (B).
  Interventions: Device: Acupuncture needles; Dietary Supplement: Soy phytoestrogens

INTERVENTIONS:
Device: Acupuncture needles — Standard acupuncture needle which is 3 cm long with diameter o.3 mm
  Arms: Acupuncture Group; Acupuncture and Soy Group
Dietary Supplement: Soy phytoestrogens — 100 millilitre of soy milk every day or 100 gram of cooked soy beans per day.
  Arms: Acupuncture and Soy Group; Soy Group

SUMMARY:
The aim of this study to determine the effect of soy phytoestrogens and acupuncture on osteoporosis in female athlete triad at adolescence age. It is hypothesized that:

- There will be no statistical significant difference between the effects of soy phytoestrogens and acupuncture on osteoporosis in female athlete triad at adolescence age. RESEARCH QUESTION: Do soy phytoestrogens and acupuncture have an effect on bone mineral density in female athlete triad at adolescence age?

DETAILED DESCRIPTION:
Many female athletes don't depend only on physical training and exercising to obtain the ideal slim and thin body. So that they follow harmful unhealthy diet to achieve the ideal body shape they are seeking. These types of diet can lead to malnutrition, menstrual disturbances, and bone loss, and these three components form a triad called female athlete triad. A limited number of studies have examined the effect of acupuncture and soy products on irregularities related to female athletes so the aim of this study is to investigate the effect of both acupuncture in line with diet modification using soy products on osteopenia in female athlete triad. Study Design: A prospective, randomized, single-blind, pre-post-test, controlled trial.

Sixty female athletes with ages ranged from 14 to 18 years, playing gymnastics and all diagnosed and referred with female athlete triad resulting in decreased bone mineral density and osteoporosis. All participants will be treated with soy products and acupuncture and will be closely followed for six months. DEXA will be used to assess bone mineral density before and after the treatment program.

ELIGIBILITY:
Inclusion Criteria:

All girls diagnosed with female athlete triad resulting in osteopenia

* Their age between 14-18 years old
* Their body mass index is less than 5 percent according to the gross motor chart
* All participants are gymnastics players
* All are medically stable
* They will be able to follow instructions

Exclusion Criteria:

* Marriage
* Pregnancy
* Taking any hormonal treatment
* Receiving any other form of traditional physical therapy modalities

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density | Six months
  DEXA(Dual-energy X-ray absorptiometry)

CONTACTS AND LOCATIONS:
Overall Officials: Hend Reda, PhD, Study Director — Badr University in Cairo
Locations (1):
- Faculty of Physical Therapy, Badr University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No